CLINICAL TRIAL: NCT03512223
Title: Intravenous and Perineural Dexamethasone for Brachial Plexus Block in Hand Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Kushelev, Assistant Professor-Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017H0244
Record Dates: First submitted 2018-04-03; First posted 2018-04-30 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Hand Surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (IV dexamethasone) (Experimental): Perineural (30ml of 0.75% ropivacaine + 0.5 ml normal saline) and IV (9.0 ml normal saline + 1 ml of 10 mg/ml Dexamethasone)
  Interventions: Drug: Dexamethasone
- Group B (IV + perineural dexamethasone) (Experimental): (IV + perineural dexamethasone): Perineural (30ml of 0.75% ropivacaine + 0.5 ml of 10 mg/ml Dexamethasone) and IV (9.5 ml normal saline + 0.5 ml of 10 mg/ml Dexamethasone)
  Interventions: Drug: Dexamethasone
- Group C (control with no adjuvant dexamethasone) (No Intervention): Perineural (30ml of 0.75 ropivacaine + 0.5 ml normal saline) and IV (10 ml normal saline)

INTERVENTIONS:
Drug: Dexamethasone — Intravenous and Perineural Dexamethasone for Brachial Plexus Block
  Arms: Group A (IV dexamethasone); Group B (IV + perineural dexamethasone)

SUMMARY:
This study aims to evaluate the if the administration of dexamethasone both around the nerve and in the vein (perineural and intravenous (IV)) will prolong the duration of pain relief from ropivacaine when compared with ropivacaine local block alone or when administered along with IV dexamethasone in patients undergoing hand surgery.

DETAILED DESCRIPTION:
This study aims to evaluate the if the administration of dexamethasone both around the nerve and in the vein (perineural and intravenous (IV)) will prolong the duration of pain relief from ropivacaine when compared with ropivacaine local block alone or when administered along with IV dexamethasone in patients undergoing hand surgery. Individuals who have hand surgery scheduled will be evaluated for eligibility in this study. Eligible and consenting patients will be randomly assigned to one of three groups (1:1:1) as follows: • Group A (IV dexamethasone): Perineural (30ml of 0.75% ropivacaine + 0.5 ml normal saline) and IV (9.0 ml normal saline + 1 ml of 10 mg/ml Dexamethasone) • Group B (IV + perineural dexamethasone): Perineural (30ml of 0.75% ropivacaine + 0.5 ml of 10 mg/ml Dexamethasone) and IV (9.5 ml normal saline + 0.5 ml of 10 mg/ml Dexamethasone) • Group C (control with no adjuvant dexamethasone): Perineural (30ml of 0.75 ropivacaine + 0.5 ml normal saline) and IV (10 ml normal saline) This study is single-blind, so the subjects will not know to which group they have been assigned. All subjects will receive at least a nerve block with a local anesthetic, or numbing agent. After written, informed consent is obtained and on the day of surgery, the research staff will collect information about the subject's medical history including allergies (seasonal and drug related), demographics (gender, age, height, weight), history of drug use, pain and nausea scores, and vital signs. All medication taken 1 month prior to treatment day will be recorded. Information will be collected from the physical examination performed by the surgeon, which is a standard procedure for the pre-operative visit, regardless of participation in the study. After being put under light sedation according to standardized sedation, as written in the protocol, one group will receive a local nerve block and numbing agent. The other two groups will receive either the nerve block and local anesthetic with intravenous dexamethasone or the nerve block and local anesthetic with both intravenous and perineural (local) dexamethasone, as described above. Details regarding the subject's surgery and anesthesia will be collected, and after your surgery, a member of the research team will provide the subject with a diary to document level of pain, movement, any episodes of nausea/vomiting, and the number of pain medicine tablets taken for up to 48 hours after surgery. The subjects will receive a follow up phone call 48 hours after the nerve block from the research team to collect the information already documented in the diary. Thus far, no evidence of dexamethasone toxicity around the nerve has been shown and no neurologic complications or infections have been reported. Only one study reported blood glucose elevations [1]. There is a potential benefit of enhancing the duration of the nerve block and therefore pain management. The results of this study will help clarify if use of dexamethasone as an adjuvant in nerve block will prolong the effect of the nerve block and reduce the heightened sensitivity to pain and burning sensation as the block wears off.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients age 18-80
* Undergoing distal radius ORIF (open reduction internal fixation) or CMC (Carpometacarpal) arthroplasty
* ASA (American Society of Anesthesiologists) I, II,III
* Patients who provide a signed written informed consent
* Have a valid phone number and be able to speak, read, and write in English

Exclusion Criteria:

* Any documented cognitive or psychological disorders that, in the opinion of the principal investigator, can interfere with the patients' pain perception
* Diabetes Mellitus
* Vulnerable populations: pregnant females, prisoners, breast feeding
* Contraindication to nerve block: local infections, bleeding disorders, shoulder deformity, allergy to local anesthetic or dexamethasone
* Severe lung disease, known contralateral phrenic nerve injury
* Previous history of chronic pain diseases requiring consistent analgesic therapy for at least 1 month prior to surgery
* Presence of any medical condition that, in the opinion of the principal investigator, should exclude the patient from the study
* BMI ≥ 40 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Duration of anesthetic blockade | 48 hours
  • The duration of anesthetic blockade measured by the time from performing the perineural block to the first reported pain at the surgical site between groups

SECONDARY OUTCOMES:
Duration of motor block | 48 hours
  • To compare the duration of motor block between groups (defined as the time between performance of the perineural block and full return of motor function in comparison to the contralateral limb)
Patient satisfaction on a scale of 0-10 (0=not satisfied at all 10=very satisfied) of pain management | 48 hours
  • To compare overall patient satisfaction of pain management between groups
48-hour postoperative units of oral morphine consumption | 48 hours
  • To compare 48-hour postoperative units of oral morphine consumption between groups
the incidence of nausea and/or vomiting within 48 hour of the block | 48 hours
  • To compare the incidence of nausea and/or vomiting within 48 hour of the block
• Rebound pain on a scale of 0-10 (0=no pain 10=worst possible pain), which is the worst level of pain experienced within the 2 hours after the block wore off | 48 hours
  • Rebound pain (the worst pain in the 2 hours after the block wore off)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kushelev, MD, Principal Investigator — Assistant Professor-Clinical
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Hussain N, Speer J, D'Souza RS, Palettas M, Abdel-Rasoul M, Uribe A, Weaver TE, Kushelev M, Coffman J, Abdallah FW. Exploring the Additive or Synergistic Effects of the Systemic and Perineural Routes of Dexamethasone as Adjuncts to Supraclavicular Block: A Randomized Controlled Trial. Anesthesiology. 2025 Jun 1;142(6):1127-1137. doi: 10.1097/ALN.0000000000005433. Epub 2025 Mar 4. PMID 40036049
- [Derived] Bei T, Liu J, Huang Q, Wu J, Zhao J. Perineural Versus Intravenous Dexamethasone for Brachial Plexus Block: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Pain Physician. 2021 Sep;24(6):E693-E707. PMID 34554686